CLINICAL TRIAL: NCT02703909
Title: A Prospective Randomized Clinical Trial Evaluating Surgical Conditions During Laparoscopic Bariatric Surgery With Deep Versus Moderate Neuromuscular Blockade
Brief Title: Surgical Conditions During Laparoscopic Bariatric Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Terri Monk, Professor, Anesthesiology, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2004620
Record Dates: First submitted 2016-02-29; First posted 2016-03-09 (Estimated); Results first posted 2018-06-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-05

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; laparoscopic surgery; neuromuscular blockade
MeSH Terms: conditions — Obesity, Morbid | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- moderate NMB + 10 mm IP (Experimental): participants will be given the muscle relaxant, rocuronium, iv to obtain a moderate neuromuscular block (NMB) which is defined as 2-3 twitches in the train of four on a neuromuscular junction monitor. The initial insufflation pressure for the laparoscopy will be 10 mm Hg pressure.
  Interventions: Drug: Rocuronium; Device: Insufflation pressure
- moderate NMB + 15 mm IP (Active Comparator): participants will be given the muscle relaxant, rocuronium, iv to obtain a moderate NMB which is defined as 2-3 twitches in the train of four on a neuromuscular junction monitor. The initial insufflation pressure for the laparoscopy will be 15 mm Hg pressure. This arm represents the usual operating conditions for this type of surgery at the University hospital.
  Interventions: Drug: Rocuronium; Device: Insufflation pressure
- deep NMB + 10 mm IP (Experimental): participants will be given the muscle relaxant, rocuronium, iv to obtain a deep NMB which is defined as 0-1 posttetanic counts on a neuromuscular junction monitor and the initial insufflating pressure will be 10 mm Hg. The initial insufflation pressure for the laparoscopy will be 10 mm Hg pressure.
  Interventions: Drug: Rocuronium; Device: Insufflation pressure
- deep NMB + 15 mm IP (Experimental): participants will be given the muscle relaxant, rocuronium, iv to obtain a deep NMB which is defined as 0-1 posttetanic counts on a neuromuscular junction monitor and the initial insufflating pressure will be 15 mm Hg. The initial insufflation pressure for the laparoscopy will be 10 mm Hg pressure.
  Interventions: Drug: Rocuronium; Device: Insufflation pressure

INTERVENTIONS:
Drug: Rocuronium — Rocuronium will be administered to achieve either a moderate (2-3 twitches) or deep (0-1 posttetanic) block depending on the group assignment
  Other Names: Zemuron
Device: Insufflation pressure — The initial insufflation pressure will be set at either 10 or 15 mm Hg depending on the group assignment
  Other Names: intra-abdominal pressure

SUMMARY:
Obesity affects more than 78 million adults in the United States and it is estimated that 35% of the US population is obese. Currently, more than 179,000 bariatric procedures are performed in the US each year with the majority of these surgeries using laparoscopic techniques. Surgeons often request deep neuromuscular blockade (NMB) during surgery, but there is no evidence that a deep NMB improves surgical conditions and that the surgeons can discriminate between a moderate and deep NMB. There is also evidence that maintaining low insufflation pressures during laparoscopic surgery may decrease postoperative pain. The goal of this prospective, randomized, assessor-blinded controlled trial is to test the hypothesis that deep NMB provides optimal surgical conditions during laparoscopic bariatric surgery in the morbidly obese patient. It will also determine if deep NMB allows the surgeon to utilize lower insufflation pressure and decreases postoperative pain requirements after laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
Subjects will be randomized to one of four groups:

1. moderate neuromuscular block (NMB) + 10 mm insufflation pressure (IP);
2. moderate NMB + 15 mm IP;
3. deep NMB + 10 mm IP; or
4. deep NMB + 15 mm IP.

A moderate NMB block will be defined as 2-3 twitches in the train of four (TOF) and a deep NMB will be defined as 0-1 posttetanic count. The surgeons will be asked to rate their satisfaction with the surgical conditions using a five-point ordinal scale ranging from 1 (extremely poor) to 5 (optimal conditions). The first rating will occur at the beginning of the procedure when the NMB level is stable at either a deep or moderate block and the intra-abdominal pressure is either 10 or 15 mm Hg (per randomization). The surgeon will be blinded to the insufflation pressure at this point. If the surgical conditions are rated as extremely poor or poor, the level of the neuromuscular block can be increased and/or the insufflation pressure can be increased to 15 mm Hg.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ASA I-III
* BMI ≥ 35

Exclusion Criteria:

* Inability to obtain written informed consent
* Pregnancy or breastfeeding
* Allergy to rocuronium, sugammadex, or any anesthetic agents used in the protocol
* Known or suspected neuromuscular disorders
* Significant renal disease with a serum creatinine ≥ 2 mg/dl f. Significant liver disease g. A family history of malignant hyperthermia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terri G Monk, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate NMB + 10 mm IP | Moderate NMB + 15 mm IP | Deep NMB + 10 mm IP | Deep NMB + 15 mm IP
Started | 36 | 37 | 36 | 35
Completed | 36 | 37 | 36 | 35
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate NMB + 10 mm IP | Moderate NMB + 15 mm IP | Deep NMB + 10 mm IP | Deep NMB + 15 mm IP | Total
Number analyzed (Participants) | 36 | 37 | 36 | 35 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (8) | 43 (11) | 50 (12) | 44 (11) | 45 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 34 | 8 | 31 | 103
  Male | 6 | 3 | 28 | 4 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 6 | 3 | 2 | 14
  White | 33 | 31 | 33 | 33 | 130
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 37 | 36 | 35 | 144

OUTCOME MEASURES:

1. Primary Outcome: Surgeon Satisfaction Scale
Description: The surgeon will grade his satisfaction with the surgical conditions using a 5 point scale with 1 - extremely poor; 2 - poor; 3 - acceptable; 4. good; 5 - optimal surgical conditions
Time Frame: day of surgery
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Moderate NMB + 10 mm IP | Moderate NMB + 15 mm IP | Deep NMB + 10 mm IP | Deep NMB + 15 mm IP
Number analyzed (Participants) | 36 | 37 | 36 | 35
Scores on a scale | 2.7 (1.0) | 4.1 (0.9) | 3.1 (1.0) | 4.6 (0.6)

2. Secondary Outcome: Number and Percentage of Subjects With Success at Low (10 mm) Insufflation Pressure
Description: The patients will be randomized to an initial insufflation pressure of 10 or 15 mm hg. If the surgeons are not satisfied with the initial operating conditions, the insufflating pressure will be increase to 15 mm Hg (if not already at that level). This will be reported as the percentage of patients who were able to have their entire surgery performed at an insufflation pressure of 10 mm Hg.
Time Frame: day of surgery
Population: The percentage of patients who were able to have their surgery completed at an IP of 10 mm
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate NMB + 10 mm IP | Moderate NMB + 15 mm IP | Deep NMB + 10 mm IP | Deep NMB + 15 mm IP
Number analyzed (Participants) | 36 | 0 | 36 | 0
Participants | 10 | 0 | 14 | 0

3. Secondary Outcome: Postoperative Opioid Requirement
Description: The participants will be given iv fentanyl or hydromorphone after surgery. They will also be given po oxycodone. The investigators will collect data on the amount of opioid that is required after surgery. This will be reported as morphine equivalents using the morphine equivalent calculator at:
Time Frame: day of surgery until hospital discharge (approximately 2-3 days)
Population: Only 24 of the patients had an IP of 10 mm throughout the surgery. The remainder of the patients either had IP of 15 mm throughout the surgery or were increased to 15 mm at the start of the surgery.
Measure: Mean (Standard Deviation); unit: morphine equivalents
Groups:
- Opioid Requirement-Subjects Who Had IP of 10 mm During Surgery: This variable reflects the amount of opioid required by the subjects in which the IP was 10 mm for the entire surgery.
- Opioid Requirement -Subjects Who Had P of 15 mm During Surgery: This variable reports the amount of opioid required in subjects who had an IP of 15 mm for the entire surgery or had their IP increase from 10 mm to 15 mm at the start of surgery.
Arm/Group | Opioid Requirement-Subjects Who Had IP of 10 mm During Surgery | Opioid Requirement -Subjects Who Had P of 15 mm During Surgery
Number analyzed (Participants) | 24 | 120
morphine equivalents | 48.8 (26.6) | 56.7 (38.6)

ADVERSE EVENTS:
Time Frame: During hospital stay approximately 3 days
Arm/Group | Moderate NMB + 10 mm IP | Moderate NMB + 15 mm IP | Deep NMB + 10 mm IP | Deep NMB + 15 mm IP
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/37 | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/37 | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 0/36 | 0/37 | 0/36 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT02703909/Prot_SAP_000.pdf